CLINICAL TRIAL: NCT01665053
Title: EVOLVE II: A Prospective Multicenter Trial to Assess the Safety and Effectiveness of the SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System (SYNERGY Stent System) for the Treatment of Atherosclerotic Lesion(s)
Brief Title: The EVOLVE II Clinical Trial To Assess the SYNERGY Stent System for the Treatment of Atherosclerotic Lesion(s)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2067; G120123 (Other: FDA)
Record Dates: First submitted 2012-08-07; First posted 2012-08-15 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug-Eluting Stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Promus Element Plus (Active Comparator): PROMUS Element Plus is a device/drug combination product composed of two components, a device (coronary stent system including a platinum chromium stent platform) and a drug product (a formulation of everolimus contained in a polymer coating).
  Interventions: Device: PROMUS Element Plus
- SYNERGY (Experimental): SYNERGY is a device/drug combination product composed of two components, a device (coronary stent system including a platinum chromium stent platform) and a drug product (a formulation of everolimus contained in a bioabsorbable polymer coating).
  Interventions: Device: SYNERGY

INTERVENTIONS:
Device: PROMUS Element Plus — A drug eluting coronary stent system
  Arms: Promus Element Plus
Device: SYNERGY — A drug eluting coronary stent system
  Arms: SYNERGY

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System for the treatment of subjects with atherosclerotic lesion(s) ≤ 34 mm in length (by visual estimate) in native coronary arteries ≥2.25 mm to ≤4.0 mm in diameter (by visual estimate).

DETAILED DESCRIPTION:
A concurrent, non-randomized, single-arm, pharmacokinetic (PK) substudy and a consecutive, non-randomized, single-arm, Diabetes substudy will also enroll under the EVOLVE II protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed
* For subjects less than 20 years of age enrolled at a Japanese site, the subject and the subject's legal representative must provide written informed consent before any study-specific tests or procedures are performed
* Subject is eligible for percutaneous coronary intervention (PCI)
* Subject has symptomatic coronary artery disease with objective evidence of ischemia or silent ischemia
* Subject is an acceptable candidate for coronary artery bypass grafting (CABG)
* Subject is willing to comply with all protocol-required follow-up evaluation

Angiographic Inclusion Criteria (visual estimate):

* Target lesion(s) must be located in a native coronary artery with a visually estimated reference vessel diameter (RVD) ≥2.25 mm and ≤4.0 mm
* Target lesion(s) length must be ≤34 mm (by visual estimate)
* Target lesion(s) must have visually estimated stenosis ≥50% and <100% with thrombolysis in Myocardial Infarction (TIMI) flow >1 and one of the following: stenosis ≥70%, abnormal fractional flow reserve (FFR), abnormal stress or imaging stress test, or elevated biomarkers prior to the procedure
* Coronary anatomy is likely to allow delivery of a study device to the target lesions(s)
* The first lesion treated must be successfully predilated/pretreated

Exclusion Criteria:

* Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation MI (STEMI)
* Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support, intractable ventricular arrhythmias, or ongoing intractable angina
* Subject has received an organ transplant or is on a waiting list for an organ transplant
* Subject is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Planned PCI (including staged procedures) or CABG after the index procedure
* Subject previously treated at any time with intravascular brachytherapy

  _ Subject has a known allergy to contrast (that cannot be adequately premedicated) and/or the trial stent system or protocol-required concomitant medications (e.g., platinum, platinum-chromium alloy, stainless steel, everolimus or structurally related compounds, polymer or individual components, all P2Y12 inhibitors, or aspirin)
* Subject has one of the following (as assessed prior to the index procedure):

  * Other serious medical illness (e.g., cancer, congestive heart failure) with estimated life expectancy of less than 24 months
  * Current problems with substance abuse (e.g., alcohol, cocaine, heroin, etc.)
  * Planned procedure that may cause non-compliance with the protocol or confound data interpretation
* Subject is receiving chronic (≥72 hours) anticoagulation therapy (i.e., heparin, coumadin) for indications other than acute coronary syndrome
* Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Subject has a white blood cell (WBC) count < 3,000 cells/mm3
* Subject has documented or suspected liver disease, including laboratory evidence of hepatitis
* Subject is on dialysis or has baseline serum creatinine level >2.0 mg/dL (177µmol/L)
* Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Subject has had a history of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
* Subject has an active peptic ulcer or active gastrointestinal (GI) bleeding
* Subject has severe symptomatic heart failure (i.e., NYHA class IV)
* Subject is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
* Subject intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* Subject with known intention to procreate within 12 months after the index procedure (women of child-bearing potential who are sexually active must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure)
* Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)

Angiographic Exclusion Criteria (visual estimate):

* Planned treatment of more than 3 lesions
* Planned treatment of lesions in more than 2 major epicardial vessels
* Planned treatment of a single lesion with more than 1 stent
* Subject has 2 target lesions in the same vessel that are separated by less than 15 mm (by visual estimate)
* Target lesion(s) is located in the left main
* Target lesion(s) is located within 3 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCx) coronary artery by visual estimate
* Target lesion(s) is located within a saphenous vein graft or an arterial graft
* Target lesion(s) will be accessed via a saphenous vein graft or arterial graft
* Target lesion(s) with a TIMI flow 0 (total occlusion) or TIMI flow 1 prior to guide wire crossing
* Target lesion(s) treated during the index procedure that involves a complex bifurcation (e.g., bifurcation lesion requiring treatment with more than 1 stent)
* Target lesion(s) is restenotic from a previous stent implantation or study stent would overlap with a previous stent
* Subject has unprotected left main coronary artery disease (>50% diameter stenosis)
* Subject has been treated with any type of PCI (i.e., balloon angioplasty, stent, cutting balloon atherectomy) within 24 hours prior to the index procedure
* Thrombus, or possible thrombus, present in the target vessel (by visual estimate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1684 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2018-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Maurer, MPH, Study Director — Boston Scientific Corporation
Locations (126):
- United States (69):
  - Baptist Medical Center - Princeton, Birmingham, Alabama
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Bakersfield Memorial Hospital, Bakersfield, California
  - University of California Davis Health System, Sacramento, California
  - Sutter Memorial Hospital, Sacramento, California
  - Alvarado Hospital Medical Center, San Diego, California
  - North Colorado Medical Center, Greeley, Colorado
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Mease Healthcare, Clearwater, Florida
  - University of Miami McKnight Brain Institute, Miami, Florida
  - MediQuest, Ocala, Florida
  - Florida Hospital Medical Center, Orlando, Florida
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - Medical Center of Central Georgia, Macon, Georgia
  - Wellstar Health Systems, Marietta, Georgia
  - Kaiser Foundation Hospital, Honolulu, Hawaii
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Prairie Cardiovascular Consultants, Ltd., Springfield, Illinois
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - St. Vincent's Medical Group, Inc., Indianapolis, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - Kings Daughters Medical Center, Ashland, Kentucky
  - Maine Medical Center, Portland, Maine
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Tufts Medical Center, Inc., Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St Mary's Duluth Clinic, Duluth, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Our Lady of Lourdes Medical Center, Haddon Heights, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - Mount Sinai - PRIME, New York, New York
  - Columbia University Medical Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Moses H. Cone Memorial Hospital-LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Rex Hospital, Raleigh, North Carolina
  - Wake Heart Research, LLC, Raleigh, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Lindner Center for Research and Education at Christ Hosp, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Sisters of Charity Providence Hospitals, Columbia, South Carolina
  - Jackson Madison County Hospital, Jackson, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - St. David's Round Rock Medical Center, Round Rock, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Henrico Doctors Hospital, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Aspirus Heart & Vascular Institute, Wausau, Wisconsin
- Australia (4):
  - The Prince Charles Hospital, Chermside, Queensland
  - Monash Medical Centre-Clayton Campus, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Austria (2):
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - AKH - Medizinische Universität Wien, Vienna
- Belgium (4):
  - Imelda Ziekenhuis, Bonheiden
  - Z.O.L - Campus St. Jan, Genk
  - UZ Leuven, Leuven
  - HHrm, Roeselare
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Hamilton Health Sciences, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Sainte-Foy, Quebec
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Finland (2):
  - University Hospital, Heart Centre, Tampere
  - Turku University Hospital, Turku
- France (8):
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest, Finistere
  - CHU de Toulouse - Hôpital Rangueil, Toulouse, Haute Garonne
  - Clinique Pasteur - Toulouse, Toulouse, Haute Garonne
  - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Bron, Rhone
  - Clinique Saint-Hilaire - Centre Frédéric Joliot, Rouen, Seine Maritime
  - Polyclinique Les Fleurs, Ollioules, Var
  - Centre Hospitalier de Lagny - Marne La Vallée, Lagny-sur-Marne
  - Hôpital Cochin, Paris
- Italy (3):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Japan (12):
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Shonan Kamakura General Hospital, Kamakura-shi, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Kyoto University Hospital, Kyoto, Kyoto
  - National Cerebral and Cardiovascular Center, Suita-shi, Osaka
  - Teikyo University Hospital, Itabashi-ku, Tokyo-To
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo-To
  - Toho University Ohashi Medical Center, Meguro-ku, Tokyo-To
  - The Cardiovascular Institute, Minatoku, Tokyo-To
  - Showa University Hospital, Shinagawa-ku, Tokyo-To
  - Department of Cardiology, Tokyo Women's Medical University, Shinjuku-ku, Tokyo-To
- P. Stradins Clinical University Hospital, Riga, Latvia
- Netherlands (3):
  - Medisch Centrum Alkmaar, Alkmaar
  - Medisch Spectrum Twente, Haaksbergerstraat, Enschede
  - St. Antonius Ziekenhuis, Nieuwegein, Nieuwegein
- New Zealand (4):
  - Ascot Angiography Ltd, Auckland
  - Middlemore Hospital, Auckland
  - North Shore Hospital, Auckland
  - Christchurch Hospital NZ, Christchurch
- Poland (3):
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - SK Przemienienia Panskiego UM im.K.Marcinkowskiego, Poznan
  - Instytut Kardiologii im.Prymasa Tysiaclecia Kardynala Stefana Wyszynskiego, Warsaw
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre, Singapore
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Derived] Kereiakes DJ, Windecker S, Jobe RL, Mehta SR, Sarembock IJ, Feldman RL, Stein B, Dubois C, Grady T, Saito S, Kimura T, Underwood P, Allocco DJ, Meredith IT. Clinical Outcomes Following Implantation of Thin-Strut, Bioabsorbable Polymer-Coated, Everolimus-Eluting SYNERGY Stents. Circ Cardiovasc Interv. 2019 Sep;12(9):e008152. doi: 10.1161/CIRCINTERVENTIONS.119.008152. Epub 2019 Aug 27. PMID 31451014
- [Derived] Kereiakes DJ, Meredith IT, Windecker S, Lee Jobe R, Mehta SR, Sarembock IJ, Feldman RL, Stein B, Dubois C, Grady T, Saito S, Kimura T, Christen T, Allocco DJ, Dawkins KD. Efficacy and safety of a novel bioabsorbable polymer-coated, everolimus-eluting coronary stent: the EVOLVE II Randomized Trial. Circ Cardiovasc Interv. 2015 Apr;8(4):e002372. doi: 10.1161/CIRCINTERVENTIONS.114.002372. PMID 25855680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1684 patients have been enrolled in the study Evolve II Randomizes Clinical trial (RCT) from 26 November 2012 until 29 Aug 2013.
  The Evolve II RCT study is anticipated to be completed (final 5-year follow-up) in 2018.
Period: Overall Study
Arm/Group | Promus Element Plus | SYNERGY
Started | 838 | 846
Completed 12-Month Clinical F/U | 797 | 822
No 12-Month F/U | 32 | 15
Death With No 12-month Clinical FU | 9 | 9
Completed | 806 | 831
Not Completed | 32 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Promus Element Plus | SYNERGY | Total
Number analyzed (Participants) | 838 | 846 | 1684
Age, Continuous [Mean (Standard Deviation); unit: yr] | 63.92 (10.50) | 63.48 (10.44) | 63.70 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 249 | 478
  Male | 609 | 597 | 1206
Race/Ethnicity, Customized [Number; unit: participants] — The Ethnicity and Race data are not mutually exclusive. For example: subject can check both "Asian" and "Native Hawaiian or other Pacific Islander", or "Caucasian" and "Hispanic or Latino".
  Therefore the sum of participants in all Categories for the Measure does not equal the Overall Number of Baseline Participants in the Arm/Group
  participants
    American Indian or Alaska native | 2 | 1 | 3
    Asian | 100 | 100 | 200
    Black,of African heritage | 37 | 52 | 89
    Caucasian | 664 | 655 | 1319
    Hispanic or Latino | 16 | 15 | 31
    Native Hawaiian or other Pacific Islander | 2 | 3 | 5
    Other | 5 | 4 | 9
    Not Disclosed | 13 | 20 | 33
Region of Enrollment [Number; unit: participants]
  Singapore | 12 | 15 | 27
  United States | 506 | 514 | 1020
  Japan | 81 | 74 | 155
  Spain | 20 | 18 | 38
  New Zealand | 13 | 11 | 24
  Canada | 56 | 58 | 114
  Latvia | 12 | 11 | 23
  Netherlands | 13 | 12 | 25
  Austria | 2 | 1 | 3
  Belgium | 50 | 50 | 100
  Finland | 14 | 16 | 30
  Denmark | 9 | 10 | 19
  Poland | 4 | 5 | 9
  Italy | 10 | 11 | 21
  Australia | 16 | 17 | 33
  France | 20 | 23 | 43
Height [Mean (Standard Deviation); unit: inches] | 67.44 (4.07) | 67.23 (4.00) | 67.33 (4.04)
Weight [Mean (Standard Deviation); unit: lbs] | 190.45 (44.29) | 190.92 (44.09) | 190.69 (44.18)
Smoking [Number; unit: participants]
  Smoking, Ever | 519 | 510 | 1029
  Smoking,Unknown | 12 | 19 | 31
  Smoking, Never | 307 | 317 | 624
Current Diabetes Mellitus [Number; unit: participants]
  Current Diabetes Mellitus | 276 | 275 | 551
  No Current Diabetes Mellitus | 562 | 571 | 1133
Hyperlipidemia Requiring Medication [Number; unit: participants]
  Hyperlipidemia Requiring Medication | 621 | 625 | 1246
  No Hyperlipidemia requiring Medication | 217 | 221 | 438
Hypertension Requiring Medication [Number; unit: participants]
  Hypertension requiring medication | 629 | 652 | 1281
  No Hypertension requiring medication | 209 | 194 | 403
History of bleeding disorder [Number; unit: participants]
  Hystory of bleeding disorder | 1 | 2 | 3
  No history of bleeding disorder | 837 | 844 | 1681
History of GI bleeding [Number; unit: participants]
  History of GI Bleeding | 0 | 2 | 2
  No History of GI Bleeding | 838 | 844 | 1682
History of Transient Ischemic Attack [Number; unit: participants]
  History of Transient Ischemic Attack | 23 | 24 | 47
  No History of Transient Ischemic Attack | 815 | 822 | 1637
History of cerebrovascular accident [Number; unit: participants]
  History of Cerebrovascular Accident | 32 | 30 | 62
  No History of Cerebrovascular Accident | 806 | 816 | 1622
History of Transient Ischemic Attack (TIA) or Cerebrovasular Accident (CVA) [Number; unit: participants]
  History of TIA or CVA | 49 | 48 | 97
  No history of TIA or CVA | 789 | 798 | 1587
History of peripheral vascular disease (PVD) [Number; unit: participants]
  History of PVD | 59 | 68 | 127
  No History of PVD | 779 | 778 | 1557
History of renal disease [Number; unit: participants]
  History of renal disease | 52 | 56 | 108
  No History of renal disease | 786 | 790 | 1576
Baseline Lesion Characteristics as determined by the Angiographic Core Laboratory, ITT Analysis Set [Number; unit: Number of lesions] — The Promus Element Plus group has 1043 lesions in 838 subjects enrolled in this treatment arm.
  The Synergy group has 1059 lesions in 846 subjects enrolled in this treatment arm.
  The measure type is number of lesions. The total number of lesions does not match with the total number of participants since some of the participants have more than one lesion.
  Number of lesions
    Left Anterior Descending (LAD) | 433 | 437 | 870
    Left Circumflex Artery (LCx) | 275 | 265 | 540
    Right Coronary Artery (RCA) | 334 | 357 | 691
    Left Main Coronary Artery (LMCA) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Target Lesion Failure (TLF) at 12 Months
Description: TLF is defined as any ischemia-driven revascularization of the target lesion, myocardial infarction (Q-wave and non-Q-wave) related to the target vessel, or cardiac death.
Time Frame: 12 months
Population: The per protocol population was used for this analysis. Therefore the number of participants analyzed is not consistent with the numbers provided in participant flow module.
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 796 | 823
percentage of participants | 6.4 | 6.4

2. Secondary Outcome: Percentage of Participants With Target Lesion Revascularization (TLR) at 12 Months.
Description: The TLR overall rate includes: TLR Percutaneous Coronary Intervention (PCI) & TLR Coronary Artery Bypass Graft (CABG).
Time Frame: 12 months
Population: Intent-to-Treat population
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 1.7 | 2.6

3. Secondary Outcome: Percentage of Participants With Target Vessel Revascularization (TVR) at 12 Months.
Description: TVR overall includes: TVR PCI & TVR CABG.
Time Frame: 12 months
Population: Intent-to- Treat
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 3.6 | 3.8

4. Secondary Outcome: Percentage of Participants With Target Vessel Failure (TVF) at 12 Month.
Description: Target Vessel Failure is defined as any ischemic-driven revascularization of the target vessel, MI related to the target vessel, or any cardiac death.
Time Frame: 12 months
Population: Intent-to-treat analysis
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 8.2 | 8.2

5. Secondary Outcome: Percentage of Participants With Myocardial Infarction at 12 Month.
Description: The MI rate includes: MI's related to the Target Vessel, MI's with unknown relationship to the Target Vessel and MI's not related to the Target Vessel.
Time Frame: 12 months
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 5.0 | 5.4

6. Secondary Outcome: Percentage of Participants With Cardiac Death at 12 Month.
Time Frame: 12 months
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 0.9 | 0.5

7. Secondary Outcome: Percentage of Participants With Non-Cardiac Death at 12 Month.
Time Frame: 12 months
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 0.2 | 0.6

8. Secondary Outcome: Percentage of Patients That Died at 12 Months.
Description: The Death rate includes Cardiac- & Non-Cardiac Death.
Time Frame: 12 months
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 1.1 | 1.1

9. Secondary Outcome: Percentage of Patients With Cardiac Death or Myocardial Infarction (MI) at 12 Month.
Time Frame: 12 months
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 5.6 | 5.6

10. Secondary Outcome: Percentage of Participants Who Died or Had an Myocardial Infarction (MI) at 12 Month.
Time Frame: 12 months
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 5.8 | 6.3

11. Secondary Outcome: Percentage of Participants Who Died, Had an Myocardial Infarction (MI) or a Target Vessel Revascularization (TVR) at12 Month.
Time Frame: 12 months
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 8.4 | 9.3

12. Secondary Outcome: Percentage of Participants With a ARC (Academic Research Consortium) Stent Thrombosis Rate at 12 Month.
Time Frame: 12 months
Population: Intent-to-treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 0.7 | 0.6

13. Secondary Outcome: Percentage of Patients With a Stroke at 12 Month.
Description: The stroke rate includes: Ischemic- , Hemorraghic- & Undetermined Stroke.
Time Frame: 12 months
Population: Intent-to-Treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 0.9 | 0.7

14. Secondary Outcome: Periprocedural Technical Success Rate.
Description: Technical Success Rate is defined as successful delivery and deployment of the study stent to the target vessel, without balloon rupture or stent embolization, and post-procedure diameter stenosis less then 30% in 2 near-orthogonal projections with TIMI 3 flow in the target lesion. Technical success is lesion based.
Time Frame: Day 1 (periprocedure)
Population: Intent-to-Treat analysis set. Promus Element Plus population: 838 subject analyzed with 1043 lesions treated with technical success achieved in 1011 lesions.
  SYNERGY population: 846 subjects analyzed with 1059 lesions treated with technical success achieved in 1041 lesions.
Measure: Number; unit: percentage of lesions
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 838 | 846
percentage of lesions | 96.9 | 98.3

15. Secondary Outcome: Periprocedural Clinical Procedural Success Rate
Description: Procedural Success Rate is defined as post-procedure diameter less then 30% in 2 near-orthogonal projections with TIMI 3 flow in all target lesions without occurrence of in-hospital cardiac death, MI, TVR. Procedural success rate is subject based.
Time Frame: Day 1 (periprocedure)
Population: Intent-to-Treat population
Measure: Number; unit: percentage of subjects
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 838 | 846
percentage of subjects | 94.3 | 94.9

16. Secondary Outcome: Percentage of Participants With a Target Lesion Failure (TLF) at 12 Month.
Time Frame: 12 month
Population: Intent-to-Treat population
Measure: Number; unit: percentage of participants
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of participants | 6.4 | 6.6

17. Secondary Outcome: Percentage of Patients With Revascularization (=All Revascularizations) at 12 Month.
Description: All CEC adjudicated revascularization at 12 month (Intent to treat population).
Time Frame: 12 Month
Population: Intent to treat population
Measure: Number; unit: percentage of patients
Arm/Group | Promus Element Plus | SYNERGY
Number analyzed (Participants) | 808 | 832
percentage of patients | 3.6 | 4.0

ADVERSE EVENTS:
Time Frame: Site-Reported Serious Adverse Events to 12 Months
Arm/Group | Promus Element Plus | SYNERGY
Serious Adverse Events (participants affected / at risk) | 262/838 | 265/846
Other Adverse Events (participants affected / at risk) | 576/838 | 567/846
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Promus Element Plus (N=838) | SYNERGY (N=846)
Cardiac disorders (Cardiac disorders) | 126 | 143
General disorders and administration site conditions (General disorders) | 49 | 45
Nervous sysytem disorders (Nervous system disorders) | 18 | 26
Injury, poisining and procedural complications (Injury, poisoning and procedural complications) | 23 | 26
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 20 | 23
Infections and infestations (Infections and infestations) | 23 | 22
Vascular disorders (Vascular disorders) | 20 | 19
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 14
Gastrointestinal disorders (Gastrointestinal disorders) | 28 | 15
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5 | 13
Renal and Urinary disorders (Renal and urinary disorders) | 15 | 14
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 11 | 14
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 7 | 8
Psychiatric disorders (Psychiatric disorders) | 4 | 6
Eye disorders (Eye disorders) | 7 | 4
Hepatobiliary disorders (Hepatobiliary disorders) | 5 | 4
Investigations (Investigations) | 5 | 4
Endocrine disorders (Endocrine disorders) | 1 | 2
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2 | 1
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 1
Immune system disorders (Immune system disorders) | 1 | 1
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1 | 0
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 0
Surgical and medical procedures (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Promus Element Plus (N=838) | SYNERGY (N=846)
Angina Pectoris (Cardiac disorders) | 104 (125) | 100 (116)
Myocardial infarction (Cardiac disorders) | 70 (70) | 74 (74)
Coronary artery dissection (Cardiac disorders) | 27 (28) | 32 (33)
Angina unstable (Cardiac disorders) | 18 (19) | 20 (24)
Acute myocardial infarction (Cardiac disorders) | 11 (12) | 17 (17)
Atrial fibrillation (Cardiac disorders) | 16 (17) | 13 (15)
Cardiac failure congestive (Cardiac disorders) | 10 (13) | 9 (10)
Bradycardia (Cardiac disorders) | 11 (11) | 8 (10)
Palpitations (Cardiac disorders) | 10 (11) | 7 (7)
Ventricular tachycardia (Cardiac disorders) | 8 (8) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 (45) | 44 (49)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 19 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 14 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 11 (11)
Dizziness (Nervous system disorders) | 27 (28) | 30 (31)
Headache (Nervous system disorders) | 21 (22) | 17 (19)
Syncope (Nervous system disorders) | 11 (11) | 13 (15)
Nausea (Gastrointestinal disorders) | 16 (16) | 12 (12)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 (11) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 5 (5)
Rectal Haemorrhage (Gastrointestinal disorders) | 9 (9) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 21 (21)
Back Pain (Musculoskeletal and connective tissue disorders) | 19 (21) | 16 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 14 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 10 (10)
Pneumonia (Infections and infestations) | 15 (15) | 17 (17)
Urinary tract infection (Infections and infestations) | 11 (12) | 10 (12)
Nasopharyngitis (Infections and infestations) | 11 (13) | 9 (10)
Contusion (Injury, poisoning and procedural complications) | 18 (18) | 12 (13)
Hypertension (Vascular disorders) | 30 (33) | 24 (25)
Hypotension (Vascular disorders) | 20 (20) | 9 (10)
Cardiac enzymes increased (Investigations) | 13 (13) | 5 (5)
Troponin increased (Investigations) | 10 (10) | 5 (5)
Haematuria (Renal and urinary disorders) | 15 (15) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 9 (11)
Drug hypersensitivity (Immune system disorders) | 14 (14) | 15 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications to public release and can embargo communications regarding trial results for a period less or equal to 45 days from the time submitted to the sponsor. If the sponsor determines the communication would be detrimental to the intellectual property, the PI will redact or modify or will refrain the publication to a publisher or other party for an additional 120 days to permit the sponsor to file patent applications or take other steps to protect interests